CLINICAL TRIAL: NCT01635400
Title: Phase Ⅱ Study of Relationship Between UGT1A1 Gene Polymorphism and Toxicity and Efficacy of Irinotecan in Small Cell Lung Cancer
Brief Title: Study of Relationship Between UGT1A1 Gene Polymorphism and Toxicity and Efficacy of Irinotecan in Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UGT1A1-01
Record Dates: First submitted 2012-06-27; First posted 2012-07-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-06

CONDITIONS: Small Cell Carcinoma of Lung
Keywords: Irinotecan; UGT1A1 Gene Polymorphisms; Small Cell Carcinoma of Lung
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- UGT1A1 wild type (6/6) (Other)
  Interventions: Drug: Irinotecan
- UGT1A1 heterozygous genotype (6/7) (Other)
  Interventions: Drug: Irinotecan
- UGT1A1 homozygous genotype(7/7) (Other)
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — irinotecan 180mg/m2 i.v. over 30 min d1,q2w

SUMMARY:
The purpose of this study is to find out the correlation between uridine diphosphate glucuronosyl transferase 1A1(UGT1A1) gene polymorphisms and the side effect and efficacy of irinotecan in patients with small cell lung cancer.

DETAILED DESCRIPTION:
In multiple studies of metastatic colorectal cancer,uridine diphosphate glucuronosyl transferase 1A1(UGT1A1) gene polymorphisms and its correlation with irinotecan-associated side effects have been confirmed.Data from several studies indicated an improved clinical outcome of patients who had received an irinotecan-based regimen.In order to find out the correlation between UGT1A1 gene polymorphisms and the side effect and efficacy of irinotecan in patients with small cell lung cancer,we designed this study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of refractory or relapsed small cell lung cancer
* Physical examination and routine laboratory tests show no contraindications to chemotherapy

Exclusion Criteria:

* Pregnant and nursing women
* Brain metastasis with symptoms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Side effect of chemotherapy | within the first 30 days (plus or minus 3 days) after chemotherapy
  myelosuppression,diarrhea

SECONDARY OUTCOMES:
response rate of chemotherapy | tumor assessments after two cycles of chemotherapy,an expected average of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yun, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China